CLINICAL TRIAL: NCT00194077
Title: Aripiprazole in Children With Symptoms of Mania
Brief Title: Study of Aripiprazole (Abilify) in Children With Symptoms of Mania
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Robert L Findling, MD, Director, Division of Child and Adolescent Psychiatry, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Children with Mania
Record Dates: First submitted 2005-09-11; First posted 2005-09-19 (Estimated); Results first posted 2013-12-05 (Estimated); Last update posted 2015-01-07 (Estimated); Status verified 2014-12

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Aripiprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aripiprazole (Active Comparator): Phase I and Phase III are open label Abilify phases where all subjects receive active Abilify
  Interventions: Drug: Aripiprazole
- Placebo (Placebo Comparator): in Phase 2 subjects are randomized to either placebo or abilify for up to 72 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aripiprazole — dosing will occur at 2mg, 5mg, 7mg, 10 mg, 12mg, or 15 mg based on weight, side effects and efficacy
  Other Names: Abilify
  Arms: Aripiprazole
Drug: Placebo — subjects in phase 2 will be randomized to active abilify or placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to look at the safety and effectiveness of aripiprazole (abilify) in children with bipolar disorder and to examine whether or not patients that respond to initial mood stabilization benefit from continued pharmacotherapy.

DETAILED DESCRIPTION:
This outpatient study will be conducted in 3 phases. Phase 1: Patients meeting entry criteria will be treated with open label aripiprazole (APZ) in order to achieve therapeutic doses of this agent. The primary objective of this phase is to stabilize the patient's mood prior to randomization in phase 2. Adjunctive treatment of attention-deficit hyperactivity disorder (ADHD) will be permitted during this phase after week 6 of phase 1. In order to be entered into Phase 2, patients must be clinically stable based on a priori criteria (see below). The maximum allowable duration of Phase 1 will be 16 weeks. Only patients who have achieved syndromal remission (not just improvement) will be eligible for randomization into phase 2.

Phase 2: Patients that achieve syndromal remission during Phase 1 will be randomized in a double-blind fashion to receive either ongoing APZ therapy or placebo therapy during Phase 2. Patients who are receiving co-administration of ADHD pharmacotherapy may continue with this during Phase 2. Patients will have an equal chance of being assigned to each of the 2 treatment arms. Randomization strata will be based on whether or not the subject is receiving ADHD pharmacotherapy and whether or not the subject is suffering from Bipolar 1 or 2 disorders. The maximum length of time a patient may remain in phase 2 will be 72 weeks. Youths who develop a major depressive episode, a manic, or mixed episode, or youths for whom continued enrollment in this phase of study is contraindicated (as determined by the patient, guardian, research team or study physician), will be withdrawn from phase 2. Youths who withdraw from phase 2 may enter Phase 3. Reason for removal from phase 2 will be documented. For those youths who successfully complete 72 weeks of participation in phase 2, trial participation will be ended. Those patients who complete phase 2 will receive follow up clinical care either at University Hospitals-Cleveland (UHC) or with a community-based physician.

Phase 3: For youths who are withdrawn during phase 2, 8-weeks of open-label treatment with APZ will be available

ELIGIBILITY:
Inclusion Criteria:

* Outpatients ages 4-9 years (inclusive)
* Patients who are anticipated to have a Young Mania Rating Scale (Young et al. 1978) of 15 or higher at baseline
* Meet DSM-IV criteria for bipolar disorder type 1 or 2, cyclothymia, or bipolar disorder not otherwise specified (BP NOS) based on the results of both a semi-structured diagnostic research assessment (K-SADS-PL supplemented with mood disorder sections from the WASH-U K-SADS) (Geller et al., 2001; Kaufman et al., 1997) and a clinical interview with a child and adolescent psychiatrist.

Exclusion Criteria:

* Patients who have a history of intolerance to APZ at doses of 0.1mg/kg/day
* Patients who have experienced a manic episode with a documented APZ dose as monotherapy treatment of 0.2 mg/kg/day
* Patients with an active neurological/medical disorder for which treatment with APZ would be contraindicated
* Patients with clinical evidence of autistic disorder, Asperger's disorder, Rett's syndrome or other pervasive developmental disorders
* Patients with clinical evidence of mental retardation
* Patients who are known to be allergic or hypersensitive to aripiprazole
* Patients who are unable to swallow pills/capsules
* Patients for whom the need for hospitalization during the course of the study appears likely
* Patients who have a general medical or neurological condition (including clinically significant abnormalities on screening laboratories) that may be considered to be the etiology of the patient's mood disorder
* Patients who have a general medical or neurological condition for which treatment with an atypical antipsychotic would be contraindicated (e.g. tardive dyskinesia)
* Patients who have a general medical or neurological condition that could interfere with the interpretation of clinical response to APZ treatment
* Patients taking psychotropic agents (other than psychostimulants) within one week of baseline (2 weeks for fluoxetine; 3 days for psychostimulants)

Ages: 4 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2004-08; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert L Findling, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- University Hospitals Case Medical Center, Cleveland, Ohio, United States

REFERENCES:
- [Result] Findling RL, Youngstrom EA, McNamara NK, Stansbrey RJ, Wynbrandt JL, Adegbite C, Rowles BM, Demeter CA, Frazier TW, Calabrese JR. Double-blind, randomized, placebo-controlled long-term maintenance study of aripiprazole in children with bipolar disorder. J Clin Psychiatry. 2012 Jan;73(1):57-63. doi: 10.4088/JCP.11m07104. Epub 2011 Nov 29. PMID 22152402
- [Derived] Findling RL, McNamara NK, Youngstrom EA, Stansbrey RJ, Frazier TW, Lingler J, Otto BD, Demeter CA, Rowles BM, Calabrese JR. An open-label study of aripiprazole in children with a bipolar disorder. J Child Adolesc Psychopharmacol. 2011 Aug;21(4):345-51. doi: 10.1089/cap.2010.0102. Epub 2011 Aug 8. PMID 21823912

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment University Hospitals, Case Medical Center
Pre-assignment Details: Open stabilization was initiated with aripiprazole at~0.1mg/kg upon phase 1, open stabilization entry, n+96. Of these, 60 subjects met priori response to advance to phase 2.
Groups:
- Aripiprazole: Random assignment with titrated dosing
- Placebo: Randomized assignment to placebo
Period: Overall Study
Arm/Group | Aripiprazole | Placebo
Started | 30 | 30
Completed | 6 (Lack of efficacy: Hypomania n=12 Cycling n=5 Mixed state=4 Mania n=1) | 0 (Lack of efficacy: hypomania n=17 Cycling n=6 Mania n=5 Mixed state n=1 Concern regarding tx n=1)
Not Completed | 24 | 30
Not completed — Lack of Efficacy | 22 | 29
Not completed — Study nonadherence | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Population: No differences.
Groups:
- Aripiprazole: Abilify (Children with Symptoms of Mania Study)
- Placebo: Placebo (Children with Symptoms of Mania Study)
- Total: Total of all reporting groups
Arm/Group | Aripiprazole | Placebo | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 30 | 30 | 60
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 7 | 18
  Male | 19 | 23 | 42
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Time in Weeks to Discontinuation
Description: Time in weeks to discontinuation due to any reason, including mood event, adverse event, or other.
Time Frame: up to 72 weeks
Measure: Mean (95% Confidence Interval); unit: time in weeks to discontinuation
Groups:
- Aripiprazole: Aripiprazole dosing dependent upon response
- Placebo: Placebo dosing to mirror active treatment
Arm/Group | Aripiprazole | Placebo
Number analyzed (Participants) | 30 | 30
time in weeks to discontinuation | 25.93 [15.08 to 36.78] | 3.00 [1.89 to 4.11]

ADVERSE EVENTS:
Arm/Group | Aripiprazole | Placebo
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

LIMITATIONS AND CAVEATS:
No deaths occured during this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes